CLINICAL TRIAL: NCT02363725
Title: Interest of COLchicine in the Treatment of Patients With Acute Myocardial INfarction and With Inflammatory Response
Acronym: COLIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9439
Record Dates: First submitted 2015-01-08; First posted 2015-02-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Inflammation; CRP; Colchicine
MeSH Terms: conditions — Inflammation | interventions — colchimax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventionnal treatment (Other): Optimal conventional treatment used for patients admitted for STEMI (ESC guidelines 2012):
  * Double anti-aggregation
  * IEC (or sartan) at best tolerated dose
  * Beta-blocker at best tolerated dose
  * High dose statin (usually atorvastatin 80 mg daily)
  * If ventricular dysfunction; inhibitor minérolcorticoïdes (the eplerenone more often)
  * Any other treatment will be logged.
  Interventions: Drug: Conventional treatment
- Conventionnal + Colchimax® (Experimental): Optimal conventional treatment + Colchimax®
  Interventions: Drug: Colchimax®; Drug: Conventional treatment

INTERVENTIONS:
Drug: Colchimax®
  Arms: Conventionnal + Colchimax®
Drug: Conventional treatment

SUMMARY:
Background:

Colchicine is an old well-known venerable drug routinely used in gout attacks for instance.

More recnetly it is regularly use in the treatment of pericarditis. It couls exert antiiflammatory effects targeting the adverse inflammation occuring incase of acute myocardial infarction, which is involved in poor outcomes or longer stay at hospital.

Endpoints:

* Main endpoint: AUC CRP during the initial hospital stay
* Secondary endpoints:

  * Clinical: oucomes
  * Imaging: ETT, MRI
  * Biological: various biomarkers

Method Randomized, controled, open-labbelled, comparing two parallel arms: conventionnal optimal treatment versus conventionnal optimal treatment + colchicine

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial inflarction (occlusion of coronary artery as assessed on the coronaro angiogram)
* Adult (18-90y)
* Men / women
* Aigned informed consent
* Health insurance

Exclusion Criteria:

* Cardiogenic shock
* Digestive troubles
* Active bowels inflammatory disease (Crhon, chronic, diarrhea...)
* Intolerance to the drug
* Renal insufficiency clearance < 30mL/min
* Immunosuppression, aplasia
* Active infectious disease, active known neoplasia, chronic inflammatory disease
* Hypersensitivity, allergy to one of studies components
* Active liver disease
* Poor hemodynamic conditions
* Recent severe sepsis
* Chronic treatment with corticoids or no steroids antiinflammatory agents
* No possibility for informed consent
* Protected by the law
* Poor abservance
* History of toxicomania, suicice attempts
* Pregnacy, breeding, project of pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
AUC CRP | 5 days

SECONDARY OUTCOMES:
Drug tolerance | 1 year
  Clinical outcome
hospitalization time | 1 year
  Clinical outcome
CRP measurement | 1 year
  Intrahospital peak CPK (Biological outcome)
CPK measurement | 1 year
  Size IDM (pic and kinetics) (Biological outcome)
Troponin-hs measurement | 1 year
  Size IDM (pic and kinetics) (Biological outcome)
Creatinine level | Day of inclusion and one month after inclusion
  Biological outcome
measurement of left ventricular end-systolic volume | Day of inclusion and one month after inclusion
  Remodeling ETT
measurement of left ventricular diastolic volume | Day of inclusion and one month after inclusion
  Remodeling ETT
measurement remodeling | One month after inclusion
  Remodeling ETT

CONTACTS AND LOCATIONS:
Overall Officials: Francois ROUBILLE, MD, PhD, Principal Investigator — University Hospital, Montpellier France
Locations (1):
- University Hospital Arnaud de Villeneuve, Montpellier, France